CLINICAL TRIAL: NCT00565487
Title: Phase I Study of Combination of Capecitabine and Erlotinib Concurrent With Radiotherapy in Patients With Non-Operable Locally Advanced Pancreatic Cancer
Brief Title: Combination Study of Capecitabine and Erlotinib Concurrent With Radiotherapy for Non-Operable Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSU 25709; OSI4058s
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Pancreatic Cancer
Keywords: Radiotherapy; Non-operable pancreatic cancer; locally advanced pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): This is a single arm dose escalation study with a cohort expansion.
  Interventions: Drug: Capecitabine, Tarceva

INTERVENTIONS:
Drug: Capecitabine, Tarceva — Capecitabine is a self-administered (oral) medication & will be dose escalated and administered in four dose levels: Level I - 600 mg/m2 bid; Level II - 700 mg/m2 bid; Level III - 825 mg/m2 bid; Level IV - 925 mg/m2 bid. Tarceva will be self-administered(orally) in an open-label, unblinded manner to all patients enrolled in the study. During the treatment period, patients will receive single agent Tarceva 100 mg/day. Treatment of Capecitabine & Tarceva is continued daily until the completeness of the radiation or toxicity.
  Other Names: Capecatine, Xeloda; Tarceva, Erlotinib, OSI-774

SUMMARY:
The primary purpose of this study is to determine the best dosage of Capecitabine and Tarceva combination in the setting of radiation and to assess treatment effectiveness, progression-free survival and overall survival.

DETAILED DESCRIPTION:
Over the past several decades, 5-fluorouracil based chemoradiation has been the cornerstone for the treatment of locally advanced non-operable pancreatic cancer. However, the survival of these patients is disappointing. The majority of the patients suffer either local progression or metastatic disease. With the availability of Capecitabine, a few pilot studies showed the the drug is convenient, tolerable and safe in combination with radiation therapy. Capecitabine demonstrated its superior anti-tumor activity with 14 months of median survival. However, these are small Phase I studies and the survival benefit needs to be further validated with larger studies. Epidermal growth factor receptor (EGFR) has been implicated in tumor growth and angiogenesis. Inhibiting EGFR by Tarceva has demonstrated effective treatment in metastatic pancreatic cancer. Anti-epidermal growth factor therapy in combination with radiotherapy has been demonstrated efficacious in other solid tumors such as head and neck cancer. We hypothesize that the combination of Tarceva and Capecitabine has synergistic anti-tumor effect. Hence, improvement of median survival could be potentially achieved with this novel combination.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of adenocarcinoma of the pancreas that is locally advanced & not amenable to resection with curative intent.
* Must not have received prior systemic therapy for locally advanced disease.
* ECOG performance status must be 0-2.
* Adequate hepatic, renal & bone marrow function.
* Radiographic evidence of disease is required.
* Life expectancy > 12 weeks.

Exclusion Criteria:

* Prior treatment with Capecitabine & other EGFR inhibitor.
* Patients with GI tract disease resulting in an inability to take oral medications.
* Significant GI disorders with diarrhea as a major symptom.
* Uncontrolled intercurrent illness including active infection,symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmias now well controlled with medication, myocardial infarction within the previous 6 months, psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with metastases.
* Patients who have had chemotherapy.
* Patients may not be receiving any other investigational agents, or have participated in any investigational drug study.
* Extensive symptomatic fibrosis of the lungs.
* Females who are pregnant or lactating.
* History of any other malignancy in the last 2 years, except prior history of in situ cancer, basal or squamous cell skin cancer are eligible.
* Known DPD deficiency.
* Receiving therapeutic doses of Coumarin-derivative anticoagulant therapy. Patients requiring anticoagulation who may be safely switched to LMWH are eligible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-12; Primary Completion 2014-08-05 (Actual); Study Completion 2014-08-05 (Actual)

PRIMARY OUTCOMES:
To determine optimal dosage for Capecitabine and Tarceva combination in the setting of radiation. | Two years

SECONDARY OUTCOMES:
To assess treatment efficacy and overall survival. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Yixing Jiang, M.D., Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States